CLINICAL TRIAL: NCT01519323
Title: An Open-label, Multicenter, Single-arm, Phase I Dose-escalation With Efficacy Tail Extension Study of Vemurafenib (RO5185426) in Pediatric Patients With Surgically Incurable and Unresectable Stage IIIC or Stage IV Melanoma Harboring BRAFV600 Mutations
Brief Title: BRIM-P: A Study of Vemurafenib in Pediatric Patients With Stage IIIC or Stage IV Melanoma Harboring BRAFV600 Mutations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to low enrollment.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO25390; 2011-000874-67 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-01-26 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vemurafenib (Experimental): Participants received vemurafenib into two separate cohorts with different starting doses based on greater than or equal to (>=)45 kilogram (kg) and other weighing less than (<)45 kg. The starting dose for participants (>=45 kg) was 720 milligram (mg) of vemurafenib by mouth twice daily (BID) and the next dose level for participants in this cohort was 960 mg by mouth BID. The starting dose level for participants weighing <45 kg was to be 480 mg of vemurafenib by mouth BID, but no participants were enrolled into this cohort.
  Interventions: Drug: vemurafenib

INTERVENTIONS:
Drug: vemurafenib — Cohort 1 (participants >=45 kg): starting dose level 720mg; next dose level 960 mg Cohort 2 (participants <45 kg): starting dose 480 mg
  Other Names: Zelboraf

SUMMARY:
This open-label, multicenter. single arm Phase I dose-escalation study with efficacy tail extension will evaluate the maximum tolerated dose/recommended dose, the safety and efficacy of vemurafenib (RO5185426) in pediatric participants (aged 12 through 17) with newly diagnosed or recurrent surgically incurable and unresectable Stage IIIC or Stage IV melanoma harboring BRAFV600 mutations. Participants will receive vemurafenib orally twice daily until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participants, 12 to 17 years of age inclusive
* Histologically confirmed surgically incurable and unresectable Stage IIIC or Stage IV (AJCC) melanoma
* Positive proto-oncogene B-Raf (BRAF) mutation result (Cobas 4800 BRAF V600 Mutation Test)
* Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Performance status: Karnofsky (for participants >/= 16 years of age) or Lansky (for participants < 16 years of age) score of >/= 60
* Adequate bone marrow, liver and renal function
* Participants must have fully recovered from the acute toxic effects of all prior therapy prior to first administration of study drug

Exclusion Criteria:

* Active or untreated central nervous system (CNS) lesions
* History of or known spinal cord compression or carcinomatous meningitis
* Anticipated or ongoing administration of anti-cancer therapies other than those administered in this study
* Previous malignancy within the past 5 years except for basal or squamous cell carcinoma of the skin, melanoma in-situ, and carcinoma in-situ of the cervix
* Previous treatment with selective/specific BRAF or Methyl Ethyl Ketone (MEK) inhibitor (previous treatment with sorafenib is allowed)
* Any previous treatment with study drug (RO5185426) or participation in a clinical trial that includes RO5185426
* Pregnant or lactating females
* Known human immunodeficiency virus (HIV) positivity or acquired immune deficiency syndrome (AIDS)-related illness, active hepatitis B virus, or active hepatitis C virus

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (8):
  - Los Angeles, California
  - Aurora, Colorado
  - Saint Petersburgh, Florida
  - Bethesda, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Memphis, Tennessee
  - Houston, Texas
- Australia (2):
  - Westmead, New South Wales
  - Brisbane, Queensland
- France (2):
  - Marseille
  - Pierre-Bénite
- Germany (3):
  - Kiel
  - Mainz
  - Tübingen
- Israel (2):
  - Jerusalem
  - Petah Tikva
- Italy (3):
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
- Wroclaw, Poland
- Bratislava, Slovakia
- Spain (2):
  - Esplugues de Llobregas, Barcelona
  - Seville, Sevilla
- United Kingdom (2):
  - Newcastle upon Tyne
  - Sutton

REFERENCES:
- [Derived] Chisholm JC, Suvada J, Dunkel IJ, Casanova M, Zhang W, Ritchie N, Choi Y, Park J, Das Thakur M, Simko S, Wan Rachel Tam N, Ferrari A. BRIM-P: A phase I, open-label, multicenter, dose-escalation study of vemurafenib in pediatric patients with surgically incurable, BRAF mutation-positive melanoma. Pediatr Blood Cancer. 2018 May;65(5):e26947. doi: 10.1002/pbc.26947. Epub 2018 Jan 19. PMID 29350463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First investigational site was activated on 22 December 2011.
Pre-assignment Details: Participants were enrolled in two separate cohorts with different starting doses based on greater than or equal to (>=)45 kilogram (kg) and other weighing less than (<)45 kg. Participants >=45 kg were then enrolled in a dose escalation period. No participants were enrolled in the <45 kg cohort.
Groups:
- Vemurafenib Dose Escalation Cohort Level 1: Participants received 720 milligram (mg) of vemurafenib by mouth twice daily (BID).
- Vemurafenib Dose Escalation Cohort Level 2: Participants received 960 mg of vemurafenib by mouth BID.
Period: Overall Study
Arm/Group | Vemurafenib Dose Escalation Cohort Level 1 | Vemurafenib Dose Escalation Cohort Level 2
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Death | 3 | 2
Not completed — Study terminated by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vemurafenib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)/Recommended Dose
Description: The MTD was defined as the dose level at which six evaluable participants had been treated and at most one participant experienced a dose limiting toxicity (DLT) and the next highest dose level was too toxic. Dose escalation occurred if 0 out of 3 or at most 1 out of 6 participant experienced DLT while being treated at a dose level; otherwise the dose was declared unsafe and thus above the MTD.
Time Frame: Up to 28 days of treatment
Population: A MTD could not be determined in this study because of the low number of participants enrolled.
Arm/Group | Vemurafenib
Number analyzed (Participants) | 0

2. Secondary Outcome: Area Under the Concentration-Time Curve for Vemurafenib
Time Frame: Pre-dose, 2, 4, 8, 12 hours post dose on Cycle 1 Day 1 and Cycle 1 Day 22 (each cycle is of 28 days)
Population: Pharmacokinetic (PK) population included all enrolled participants who received at least one dose or a partial dose of study treatment and provided at least one post-dose blood sample for PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per millitre (h*ng/mL)
Groups:
- Vemurafenib 720 mg: Participants enrolled in the first cohort received vemurafenib 720 mg by mouth BID.
- Vemurafenib 960 mg: Participants enrolled in the second cohort received vemurafenib 960 mg by mouth BID.
Arm/Group | Vemurafenib 720 mg | Vemurafenib 960 mg
Number analyzed (Participants) | 3 | 3
hour*nanogram per millitre (h*ng/mL)
  Cycle 1 Day 1 | 16300 (80.5) | 57000 (95.5)
  Cycle 1 Day 22 | 486000 (26.7) | 963000 (23.4)

3. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which did not necessarily have to have a causal relationship with study treatment.
Time Frame: Up to approximately 2 years 11 months
Population: Safety population included all participants who received at least one dose or a partial dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 6
participants | 6

4. Secondary Outcome: Best Overall Response Rate (BORR)
Description: BORR was assessed by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. BORR was defined as the number of participants who achieved a complete response (CR) or partial response (PR). CR was defined as complete disappearance of all target lesions and non-target disease. PR was defined as a >=30% decrease under baseline of the sum of diameters of all target lesions. BORR was summarized along with the associated exact 95% confidence interval (CI) using the method of Clopper-Pearson.
Time Frame: Up to 2 years
Population: Intent to treat population included all participants enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 6
percentage of participants | 0 [0 to 45.93]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the number of participants that achieved a CR, PR or stable disease (SD) (SD for at least 6 weeks) as assessed by investigators according to the RECIST v1.1. CR was defined as complete disappearance of all target lesions and non-target disease. PR was defined as at >=30% decrease under baseline of the sum of diameters of all target lesions. SD was defined as steady state of disease with neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
Time Frame: Up to 2 years
Population: Intent to treat population included all participants enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 6
percentage of participants | 66.7

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time between the day of first treatment and the first documentation of progressive disease or death. Progression was defined as a 20% increase in the sum of the longest diameter of target lesions, the appearance of new lesions and increase of at least 5 mm in the sum of diameters of target lesions. Participants who were withdrawn from the study without documented progression were to be censored at the date of the last known tumor assessment when the participant was known to be progression free. Median PFS was estimated using Kaplan-Meier method and 95% CI for median was computed using the Brookmeyer and Crowley method.
Time Frame: Randomization date of first subject until disease progression or death or which ever occur first (2 years)
Population: Intent to treat population included all participants enrolled.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vemurafenib
Number analyzed (Participants) | 6
days | 134.5 [83.0 to 157.0]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time between the date of first treatment to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of their last being known alive. Median overall survival was estimated using Kaplan-Meier method and 95% CI for median was computed using the Brookmeyer and Crowley method.
Time Frame: Randomization date of first subject until death (2 years)
Population: Intent to treat population included all participants enrolled.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vemurafenib
Number analyzed (Participants) | 6
days | 246.5 [156.0 to 364.0]

ADVERSE EVENTS:
Time Frame: All AEs were reported for approximately 2 years 11 months. Related serious adverse events were required to be reported regardless of the time elapsed from the last study drug administration, even if the study had been closed.
Description: An AE was defined as any untoward medical occurrence in a participant administered the investigational product which does not necessarily have a causal relationship with this treatment.
Arm/Group | Vemurafenib
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=6)
Adrenal insufficiency (Endocrine disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=6)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 3
Chest pain (General disorders) | 1
Influenza like illness (General disorders) | 1
Pain (General disorders) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Scrotal abscess (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood phosphorus increased (Investigations) | 1
Carbon dioxide decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Haemoglobinuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hot flush (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Hypothyroidism (Endocrine disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated on 18 December 2015 by the Sponsor due to recruitment challenges and therefore low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.